CLINICAL TRIAL: NCT04950166
Title: A Phase 2, Open-Label Study to Evaluate the Performance and Safety of ONM100, an Intraoperative Fluor Imaging Agent for the Detection of Peritoneal Mets
Brief Title: A Study to Evaluate ONM100, an Intraoperative Fluor Imaging Agent for the Detection of Peri Mets
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OncoNano Medicine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ON-1003
Record Dates: First submitted 2021-06-25; First posted 2021-07-06 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Peritoneal Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms

STUDY DESIGN:
Intervention Model Description: A two group interventional, open-label, single arm trial where each patient is his/her own intrapatient control. All patients will receive a single dose of pegsitacianine administered intravenously prior to standard of care surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fluorescence imaging with pegsitacianine (Experimental): 1 mg/kg of pegsitacianine administered IV 24-72 hours prior to surgery.
  Interventions: Drug: pegsitacianine

INTERVENTIONS:
Drug: pegsitacianine — An intraoperative nanoparticle-based fluorescence imaging agent comprised of micelles covalently conjugated to indocyanine green (ICG).
  Other Names: ONM-100

SUMMARY:
Peritoneal carcinomatosis (PC) results from the metastasis of a primary cancer of the peritoneum (e.g., appendiceal, ovarian, uterine, colorectal, and gastric cancers) that then disseminates throughout the abdominal cavity. Historically progression to PC was considered terminal and resulted in survival times on the scale of a few months with palliative care being the best option for patients. More recently, cytoreductive surgery (CS) has emerged as a means to prolong and improve patient lives with a median increase in survival of up to ~5 years. It has been reported that for every 10% increase in cytoreduction there is a 5.5% increase in median survival time. In addition to surgical tumor debulking within the peritoneal space, it has also been shown that coupling surgical intervention with hyperthermic intraperitoneal chemotherapy (HIPEC) can have an even greater impact on patient outcomes. Pegsitacianine, a micellar fluorescence agent, exploits the ubiquitous pH differences observed between cancerous and normal tissues. This in turn, provides a highly sensitive and specific fluorescence response after localizing within the tumor microenvironment, thus allowing the detection of primary tumors, their margins, metastatic disease, and tumor-containing lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* Imaging and biopsy confirmed metastatic disease of peritoneal origin

Exclusion Criteria:

* Known hypersensitivity or allergy to any component of pegsitacianine
* Tumor locations the surgeon deems unfeasible to image intraoperatively
* Excessive and/or generalized metastatic disease deemed inoperative by the surgeon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2023-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wagner, MD, Principal Investigator — Allegheny Health Network
Locations (5):
- United States (5):
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical Center / James Cancer Hospital, Columbus, Ohio
  - Perelman School of Medicine, University of Pennsylvania, Philadelphia, Pennsylvania
  - AHN Cancer Institute, West Penn Hospital, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients scheduled for cytoreductive surgery of the peritoneum were eligible for enrollment into the study at major oncologic surgical centers. The trial opened to enrollment in September 2021 with the first patient consenting Nov 30, 2021.
Period: Overall Study
Arm/Group | Fluorescence Imaging With Pegsitacianine
Started (51 patients consented; however, 1 patient withdrew consent prior to dosing.) | 51
Completed (All patients completed as intent-to-treat) | 50
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All subjects who received >75% of the intended dose of pegsitacianine, had a minimum of 1 image collected during their procedure, and had the opportunity for post-SOC evaluation of the thoracic cavity.
Arm/Group | Fluorescence Imaging With Pegsitacianine
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 59 [27 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 35
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients That Had at Least One Additional Lesion Detected Under Pegsitacianine Guidance Following CRS That Was Confirmed as Positive for Disease by Pathological Evaluation
Description: Percentage of patients that had at least one additional lesion detected under pegsitacianine guidance following standard of care cytoreductive surgery that would have been left behind had imaging not been performed and was confirmed to be positive for disease by pathological evaluation.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Fluorescence Imaging With Pegsitacianine
Number analyzed (Participants) | 40
Participants | 20

2. Secondary Outcome: Sensitivity of Pegsitacianine at Detecting Presence of Tumor Within the Tissue Specimen
Description: # of true positive specimens divided by the (#of true positive specimens + # of false negative specimens)
Time Frame: 7 days
Population: 282/359 specimens were collected
Measure: Number (95% Confidence Interval); unit: ratio
Units Other Than Participants: tissue specimens
Arm/Group | Fluorescence Imaging With Pegsitacianine
Number analyzed (Participants) | 40
Number analyzed (tissue specimens) | 359
ratio | .786 [.7 to .866]

3. Secondary Outcome: Specificity of Pegsitacianine at Detecting Presence of Tumor Within the Tissue Specimen
Description: # of True Negative Specimens divided by the (# of True Negative Specimens + # of False Positive Specimens)
Time Frame: 7 days
Population: 164/291 specimens collected
Measure: Number (95% Confidence Interval); unit: ratio
Units Other Than Participants: tissue specimens
Arm/Group | Fluorescence Imaging With Pegsitacianine
Number analyzed (Participants) | 40
Number analyzed (tissue specimens) | 291
ratio | .564 [.481 to .655]

4. Secondary Outcome: Negative Predictive Value of Pegsitacianine
Description: # of True negative specimens divided by the (# of true negative specimens + # of false negative specimens)
Time Frame: 7 days
Population: 164/241 specimens collected
Measure: Number (95% Confidence Interval); unit: ratio
Units Other Than Participants: tissue specimens
Arm/Group | Fluorescence Imaging With Pegsitacianine
Number analyzed (Participants) | 40
Number analyzed (tissue specimens) | 241
ratio | .68 [.566 to .797]

5. Secondary Outcome: Positive Predictive Value of Pegsitacianine
Description: # of true positive specimens divided by the (# of true positive + # of false positive specimens)
Time Frame: 7 days
Population: 282/409 specimens collected
Measure: Number (95% Confidence Interval); unit: ratio
Units Other Than Participants: tissue specimens
Arm/Group | Fluorescence Imaging With Pegsitacianine
Number analyzed (Participants) | 40
Number analyzed (tissue specimens) | 409
ratio | .689 [.595 to .780]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for ~2 months. Starting from time of single dose infusion (24-72 hours prior to surgery) through the 28 day visit following hospital discharge.
Arm/Group | Fluorescence Imaging With Pegsitacianine
All-Cause Mortality (participants affected / at risk) | 2/50
Serious Adverse Events (participants affected / at risk) | 17/50
Other Adverse Events (participants affected / at risk) | 17/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluorescence Imaging With Pegsitacianine (N=50)
Sepsis (Infections and infestations) | 3 (3) — Complication related to surgery (Not related to pegsitacianine)
Device Dislocation (Product Issues) | 1 (1) — right ureteral stent migration occurred as a result of the surgical procedure
Abdominal Infection (Infections and infestations) | 2 (2)
Wound Abscess (Infections and infestations) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) — fatal
Gastric Perforation (Gastrointestinal disorders) | 1 (1)
Large Intestine Perforation (Gastrointestinal disorders) | 1 (1)
Ileal Perforation (Gastrointestinal disorders) | 1 (1)
Intra-abdominal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Embolism (Vascular disorders) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1)
Multiple Organ Dysfunction Syndrome (General disorders) | 1 (1) — fatal
Device Dislocation (Product Issues) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluorescence Imaging With Pegsitacianine (N=50)
Infusion Related Reactions (Injury, poisoning and procedural complications) | 14 (14) — mild to moderate and self-limiting
Alanine Aminotransferase Increased (Investigations) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 2 (2)
Blood Lactate Dehydrogenase Increased (Investigations) | 2 (2)

LIMITATIONS AND CAVEATS:
Trial patients served as their own control since near infrared imaging was withheld until primary completion of surgery, which was defined by the surgeon.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT04950166/Prot_002.pdf
  • Statistical Analysis Plan (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT04950166/SAP_003.pdf